CLINICAL TRIAL: NCT04134793
Title: Correlation of Atrial Fibrillation Recurrence After Bipolar Radiofrequency Ablation With microRNA Expression
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Principal Investigator, Jian Zhao, associate professor, Henan Institute of Cardiovascular Epidemiology
Other Study IDs: HenanICE201901
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation, ablation, microRNA
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — microRNA from left atrium appendage
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sinus group: Six-month follow-up, by holter ECG record，the patients keep normal sinus after atrial fibrillation radiofrequency ablation.
  Interventions: Procedure: radiofrequency ablation
- atrial fibrillation recurrence group: Six-month follow-up, by holter ECG record，the patients again suffer from atrial fibrillation after atrial fibrillation radiofrequency ablation.
  Interventions: Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: radiofrequency ablation — bipolar radiofrequency ablation by ablation forceps

SUMMARY:
The recurrence rate of atrial fibrillation (AF) after bipolar radiofrequency ablation was about 30%. Besides the factors, left atrium diameter, the duration of AF, NT-proBNP, and ejection fraction(EF), some studies demonstrated that the specific microRNA expression (miRNA1, miRNA19,miRNA23, miRNA409 ) showed the significant change in AF patients compared with normal sinus patients, who underwent catheter ablation. Therefore, the correlation of atrial fibrillation recurrence and above-mentioned microRNA after bipolar radiofrequency ablation remained unclear, although bipolar radiofrequency ablation had high rate of sinus.

DETAILED DESCRIPTION:
Numerous studies identify specific microRNA (miRNA) expression profiles associated with atrial fibrillation (AF), changes in plasmamiRNA expression in pre-and post-operativeAFpatients who have received catheterisation . The correlation of atrial fibrillation recurrence and above-mentioned microRNA after bipolar radiofrequency ablation remain poorly characterized.

This study aimed to reveal disease-related biomarkers by detecting plasmamiRNA expression in AF patients, and examining the levels of AF-specific miRNAs in patients after bipolar radiofrequency ablation, in order to help gauge therapeutic effects and assess prognosis.

A total of 50 Han Chinese patients with AF who had received bipolar radiofrequency ablation recruited to the study. Atrial fibrillation-specific plasma miRNAs were detected by sequencing and quantitative reverse transcription polymerase chain reaction. According to AF recurrence rate of about 30%, the expression levels of AF-specific miRNAs were investigated in15 post-operative AF patients and 35 patients with normal sinus after ablation,to explore changes in miRNA expression.

ELIGIBILITY:
Inclusion Criteria:

persistent atrial fibrillation, with alone mitral valve stenosis or regurgitation

Exclusion Criteria:

left atrium more than 60mm ejection fraction less than 30% complicated with other valve disease of aortic valve stenosis or regurgitation

Ages: 14 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Study Population include persistent atrial fibrillation with mitral valve stenosis or regurgitation alone. Surgery procedure is mitral valve repair or replacement. Left atrium appendage was harvested for later tissue miRNA study. Six-month follow-up was performed by holter and echocardiography.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
atrial fibrillation recurrence rate | six months after bipolar radiofrequency ablation
  Holter ECG record
miRNA expression difference | six months after bipolar radiofrequency ablation
  miRNA-1, miRNA-19, miRNA-23, miRNA-29,miRNA-409,

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqiang Quan, doctor, Study Director — Henan Provincial People' Hospital
Locations (1):
- Henan Provincial People' Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sardu C, Santamaria M, Paolisso G, Marfella R. microRNA expression changes after atrial fibrillation catheter ablation. Pharmacogenomics. 2015 Nov;16(16):1863-77. doi: 10.2217/pgs.15.117. Epub 2015 Nov 10. PMID 26554530
- [Background] Philpott JM, Zemlin CW, Cox JL, Stirling M, Mack M, Hooker RL, Morris A, Heimansohn DA, Longoria J, Gandhi DB, McCarthy PM. The ABLATE Trial: Safety and Efficacy of Cox Maze-IV Using a Bipolar Radiofrequency Ablation System. Ann Thorac Surg. 2015 Nov;100(5):1541-6; discussion 1547-8. doi: 10.1016/j.athoracsur.2015.07.006. Epub 2015 Sep 19. PMID 26387721
- [Background] Gal P, Marrouche NF. Magnetic resonance imaging of atrial fibrosis: redefining atrial fibrillation to a syndrome. Eur Heart J. 2017 Jan 1;38(1):14-19. doi: 10.1093/eurheartj/ehv514. Epub 2015 Sep 25. PMID 26409008
- [Background] Briasoulis A, Sharma S, Telila T, Mallikethi-Reddy S, Papageorgiou N, Oikonomou E, Tousoulis D. MicroRNAs in Atrial Fibrillation. Curr Med Chem. 2019;26(5):855-863. doi: 10.2174/0929867324666170920151024. PMID 28933293
- [Background] McManus DD, Tanriverdi K, Lin H, Esa N, Kinno M, Mandapati D, Tam S, Okike ON, Ellinor PT, Keaney JF Jr, Donahue JK, Benjamin EJ, Freedman JE. Plasma microRNAs are associated with atrial fibrillation and change after catheter ablation (the miRhythm study). Heart Rhythm. 2015 Jan;12(1):3-10. doi: 10.1016/j.hrthm.2014.09.050. Epub 2014 Oct 9. PMID 25257092
- [Background] van den Berg NWE, Kawasaki M, Berger WR, Neefs J, Meulendijks E, Tijsen AJ, de Groot JR. MicroRNAs in Atrial Fibrillation: from Expression Signatures to Functional Implications. Cardiovasc Drugs Ther. 2017 Jun;31(3):345-365. doi: 10.1007/s10557-017-6736-z. PMID 28752208
- [Background] Liu T, Zhong S, Rao F, Xue Y, Qi Z, Wu S. Catheter ablation restores decreased plasma miR-409-3p and miR-432 in atrial fibrillation patients. Europace. 2016 Jan;18(1):92-9. doi: 10.1093/europace/euu366. Epub 2015 Mar 16. PMID 25782451
- [Background] Wang M, Sun L, Ding W, Cai S, Zhao Q. Ablation alleviates atrial fibrillation by regulating the signaling pathways of endothelial nitric oxide synthase/nitric oxide via miR-155-5p and miR-24-3p. J Cell Biochem. 2019 Mar;120(3):4451-4462. doi: 10.1002/jcb.27733. Epub 2018 Oct 9. PMID 30302809
- [Background] Jia X, Zheng S, Xie X, Zhang Y, Wang W, Wang Z, Zhang Y, Wang J, Gao M, Hou Y. MicroRNA-1 accelerates the shortening of atrial effective refractory period by regulating KCNE1 and KCNB2 expression: an atrial tachypacing rabbit model. PLoS One. 2013 Dec 30;8(12):e85639. doi: 10.1371/journal.pone.0085639. eCollection 2013. PMID 24386485